CLINICAL TRIAL: NCT06705231
Title: Does Deciding Not to Participate in a Lifestyle Intervention Affect the Long-term Change in Psychosocial Well-being for Children With Obesity?
Brief Title: Childhood Obesity, Decided Not to Participate, Lifestyle Intervention and Psychosocial Well-being.
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus Municipality, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 3662
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Obesity; Psychosocial Well-being
Keywords: Decided not to Participate; Lifestyle Intervention; Pediatric Obesity; Psychosocial Well-being; Long-term impact
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Decided not participate group: Children aged 5-10 years with obesity from the city of Aarhus, who decided not to participate in the lifestyle intervention in Aarhus municipality.
  Interventions: Behavioral: The Aarhus-intervention
- Intervention group: Children aged 5-10 years with obesity who participated in a one-year lifestyle intervention in Aarhus municipality.
  Interventions: Behavioral: The Aarhus-intervention
- Non-intervention group: Children aged 5-10 years with obesity from the city of Aarhus, who were never invited to participate in the intervention.

INTERVENTIONS:
Behavioral: The Aarhus-intervention — A multifactorial family-centered lifestyle intervention with a maximum duration of one year, corresponding to three-four visits. Participants were offered complimentary weekly supervised physical activity. The day-to-day intervention was managed by specialized nurses at local healthcare centers, at the participants' homes, or in a local clinic.
  Groups: Decided not participate group; Intervention group

SUMMARY:
Childhood obesity has been associated with an increased risk of impaired psychosocial well-being and the development of depression and anxiety. However, little is known about the long-term psychosocial impact on children with obesity who decided not to participate in lifestyle interventions, representing a critical gap in literature.

This study includes approximately 400 children with obesity aged 5-10 years living in Aarhus municipality in the time-period 2014-2020, who either decided not to participate in a lifestyle intervention, were not invited to participate or attended the intervention. During that period the children annually completed the Danish National Well-being Questionnaire (DNWQ) in school. The DNWQ is a national questionnaire used to examine the well-being and learning environment in Danish schoolchildren.

The aim of this study is to investigate the long-term impact on psychosocial well-being for children with obesity deciding not to participate in a family-centered lifestyle intervention compared to children who attended the intervention, and to children never invited to participate in the intervention. The study will combine data from mandatory health check-ups at school, the Danish National Registries, and the Danish agency for IT and Learning (STIL), The ministry of Education.

DETAILED DESCRIPTION:
Childhood obesity is increasing worldwide and is associated with an increased risk of developing non-communicable lifestyle diseases later in life, while reduced psychosocial well-being often occurs during childhood. Children living with obesity suffer from poor self-esteem, which have been associated with increased levels of sadness and loneliness. They also experience a higher degree of bullying, have lower quality of life, and a greater risk of depression as compared to their peers living without obesity. Family-centered lifestyle interventions using a multifactorial approach are still considered the first line treatment for addressing childhood obesity. The literature suggests that this type of intervention can stabilize or to some extent reduce weight when treating children with obesity. In addition, various studies have reported positive effects of obesity interventions on psychosocial well-being in children and adolescents.

Previous studies have reported life stressors, societal norms of weight and body size, as well as earlier experiences with the health care system to be the primary determinants for caregivers not letting their children with obesity participate in lifestyle interventions. However, no studies have been able to describe if deciding not to participate in a lifestyle intervention affects the psychosocial well-being in children with obesity.

The aim of this study is therefore to investigate the long-term impact on psychosocial well-being for children with obesity deciding not to participate in a family-centered lifestyle intervention (decided not to participate group) compared to children who attended the intervention (intervention group), and to children never invited to participate in the intervention (non-intervention group). As a secondary objective, we aim to investigate the effect that is not caused by the weight change by adjusting for this.

Study design: This observational cohort study will combine data from mandatory health examinations at school, the Danish National Registries, and the Ministry of Education for children with obesity living in Aarhus municipality, Denmark between August 1st, 2014, and June 30th, 2020. The last possible day of follow-up will be February 1st, 2023.

The participants:

This study will include children aged 5-10 years with obesity living in Aarhus municipality, who either decided not to participate in a lifestyle intervention in Aarhus (decided not to participate group), were not invited to participate (non-intervention group), or attended the intervention (intervention group). The inclusion visit will be defined as the day of deciding not to participate in the intervention (decided not to participate group), the first day of attending the intervention (intervention group), or the first observation with obesity (non-intervention group).

Obesity will be defined by the International Obesity Task Force (IOTF) guideline as an iso-BMI >= 30 kg/m2 adjusted for age and sex.

This trial will include:

* Approximately 70 children with obesity deciding not to participate in the intervention (decided not to participate group)
* Approximately 110 children with obesity treated with the one-year lifestyle intervention (intervention group)
* Approximately 230 children with obesity who were not invited to participate in the intervention (non-intervention group)

Data-collection and analyses:

Children who attended, decided not to participate, or were never invited to participate in the intervention will be identified using data from TM-Sund. Data recorded at health check-ups at the school containing height and weight will also be extracted from TM-Sund. TM-Sund is a data capturing tool used by the community health care nurses employed at Aarhus municipality.

The DNWQ data will be obtained from the Danish agency for IT and Learning (STIL), The ministry of Education.

Data on socioeconomic status (SES), immigration, family structure, and psychiatric diagnoses will be obtained from the National Danish Registers through Statistics Denmark.

Ethics & Permissions:

The local committee on health ethics have approved the overall project and data transfer (rec.no 1-45-70-27-20). The project is internally reported to the University of Aarhus (rec no. 3662). The project has achieved approval from The Danish Data Protection Agency and the Principal Investigator has been granted access to data from registers from Danish Statistics.

The researchers have no conflict of interest to declare.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion visit between August 1st, 2014, and June 30th, 2020.
* Obesity at time of referral as defined by the IOTF guideline as an iso-BMI >= 30 kg/m2 adjusted for age and sex.
* Age between 5 and 10 years at inclusion visit.
* A measure of weight and height within 6 months before or after time of inclusion
* A completed DNWQ at inclusion:

  * The decided not to participate / non-intervention groups - with a timeframe between 6 months prior to and 6 months after inclusion.
  * The intervention group - with a timeframe between 10 months prior to and 2 months after inclusion.
* A completed DNWQ at follow-up (1 to 3 years after inclusion visit).

Exclusion Criteria:

• Children first decided not to participate, but subsequently accepting the intervention.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with obesity, 5-10 years of age living in Aarhus municipality between August 1st, 2014, and June 30th, 2020. The children have either received treatment with a one-year multifactorial family-centered lifestyle intervention, decided not to participate in the intervention or where never invited to participate in the intervention.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Change in psychosocial well-being as assessed by the DNWQ, obtained from the Danish agency for IT and Learning (STIL), The ministry of Education. | Time Frame: Annually from August 1st, 2014, to February 1st, 2023
  The impact on psychosocial well-being will be assessed with responses to specific items regarding psychosocial well-being related to school from the DNWQ at time of inclusion and at follow-up. At follow-up, we will prioritize completed questionnaires closest to two years from time of inclusion visit.
  The DNWQ is a national questionnaire completed annually in primary school and used to examine how primary schoolchildren perceive their well-being and learning environment in school.
  The following psychosocial well-being items have been selected:
  1. Question:
     Are you happy with your school?
  2. Questions:
     Do you feel lonely at school?
  3. Question:
     Have you been bullied this school year?
  4. Question:
     Does your stomach ache when you are at school?
  5. Question:
     Are you good at solving your problems?
  6. Question:
     Can you concentrate during class?
  7. Question:
  Are you good at helping each other in class?

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Aarhus, Arhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Participant data (IPD) will be available on reasonable request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT06705231/Prot_SAP_000.pdf